CLINICAL TRIAL: NCT06542887
Title: Efficacy and Safety of Black Seed Oil as Adjunctive Therapy in Pediatrics With Attention-Deficit/Hyperactivity Disorder
Brief Title: Black Seed Oil in ADHD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Manar Hosney, Clinical Pharmacist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BHCL463
Record Dates: First submitted 2024-08-03; First posted 2024-08-07 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: ADHD
Keywords: ADHD, Atomoxetine, Oxidative stress, Neuroinflammation, Antioxidants, Nigella sativa, Vanderbilt Assessment Scale, Quality of life, CHQ-PF28
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neuroinflammatory Diseases | interventions — Atomoxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Open labeled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black Seed Oil Group (Experimental)
  Interventions: Drug: Atomoxetine; Drug: Black Seed Oil Cap/Tab
- Controlled Group (Active Comparator)
  Interventions: Drug: Atomoxetine

INTERVENTIONS:
Drug: Atomoxetine — Participants will continue receiving their treatment with atomoxetine at a dose of 0.5-1.4 mg/kg/day
Drug: Black Seed Oil Cap/Tab — Participants will receive black seed oil in the form of soft gelatin capsule 450 mg at a dose of 40-80 mg/kg/day given in one to two divided doses after meals for 12 weeks.
  Arms: Black Seed Oil Group

SUMMARY:
Attention-Deficit/Hyperactivity Disorder is one of the most prevalent neuropsychiatric disorders affecting children with known persistence into adulthood in about 60% of patients. The mainstay treatment for ADHD is the pharmacological treatment involving stimulants (methylphenidate, amphetamines) and non-stimulants (atomoxetine, guanfacine, clonidine). Although these options have been found to be effective, these agents may not always be promising, as a proportion of patients may not respond or may not be able to tolerate their adverse events. Thus, increasing studies are exploring alternative therapies for ADHD, focusing on the neuroprotective effects of dietary and natural compounds like antioxidants that can be serving as an alternative or supplement to classical treatment with fewer side effects. Oxidative stress and neuroinflammation have been extensively addressed in ADHD and several studies on antioxidants in pediatrics with ADHD have shown promising results in improving symptoms and reducing scores on ADHD questionnaires.

Black seed oil (BSO) has shown anti-inflammatory and antioxidant properties in several human studies. Also numerous in-vitro studies have shown that nigella sativa possesses neuroprotective effects that are attributed to its antioxidant and anti-inflammatory effects. Thymoquinone (TQ) possesses the majority of nigella sativa oil (NSO) therapeutic benefits with the ability to target the central nervous system owing to its low molecular weight and lipophilic nature. In rats, thymoquinone administration significantly improved cognition by enhancing cholinergic function, synaptic plasticity, and attenuating oxidative damage and neuroinflammation, as shown by increased SOD and TAC and reduced MDA, NO, TNF-α immunoreactivity, and AChE activities. Previous human studies suggested that nigella sativa can stabilize mood, reduce anxiety, and regulate cognition, attention, and memory. In a previous animal study on ADHD mice model, Nigella sativa oil showed a reduction in inattention and hyperactivity with lower glutamate levels, and also showed higher recognition memory, glutathione peroxidase levels, dopamine levels, and neuronal density compared to the ethanol group only.

DETAILED DESCRIPTION:
Attention-Deficit/Hyperactivity Disorder (ADHD) is a childhood-onset neurodevelopmental disorder characterized by age-inappropriate levels of inattention and hyperactivity/impulsivity symptoms that interfere with functioning or development. Based on the predominant symptoms, the Diagnostic and Statistical Manual of Mental Disorders-Fifth Edition (DSM-V) classifies ADHD into three subtypes: predominantly inattentive (ADHD-I), predominantly hyperactive/impulsive (ADHD-H), and combined (ADHD-C). To be categorized into one of those subtypes, the diagnostic criteria for ADHD in children requires the presence of six out of nine specified symptoms in either the inattentive or hyperactive/impulsive domains, or both, persisted for at least 6 months prior to the age of 12 and caused impairment in at least two settings. Children and adolescents with ADHD face difficult formative years due to their impulsive behavior and slower rates of processing information, leading to poor performance on exams, lower grades, and higher school dropout rates. In addition, their low self-esteem leads to problems in social relationships and a tendency for substance abuse. This disorder often presents with one or more comorbidities such as anxiety disorders, oppositional defiant disorder, conduct disorder, and major depressive disorder, leading to extra challenges for them.

Attention-Deficit/Hyperactivity Disorder is one of the most prevalent neuropsychiatric disorders affecting children with known persistence into adulthood in about 60% of patients. A meta-analysis of 175 studies worldwide revealed that ADHD prevalence in children and adolescents is 7.2%. In Africa, the prevalence of ADHD in children and adolescents was 7.47%. In Egypt, ADHD prevalence among adolescents has reached as high as 9.4%. The diagnosis of ADHD in boys is approximately double that of girls.

The exact etiology and risk factors for ADHD remain unknown. However, studies showed that multiple genetic and environmental factors interact during early development to create a neurobiological susceptibility to this multifactorial disorder. The pathophysiology related to ADHD is associated with brain abnormalities that lead to cognitive and functional deficits. This disorder extensively addresses a deficit in specific brain regions, primarily the prefrontal cortex (PFC), caudate, and cerebellum together with their linking networks, the dopaminergic and noradrenergic systems, that regulate attention, thoughts, emotions, behavior, and actions.

Oxidative stress (OS) and neuroinflammation along with their role in brain dysfunction have been extensively addressed in ADHD. Brain is particularly susceptible to OS because of its high metabolic rate, high oxygen utilization, high lipid contents, and relatively low antioxidant concentration. A previous study in children with ADHD reported an impairment in serum oxidant/antioxidant balance reflected by lower ratios of serum nitric oxide/melatonin and serum malondialdehyde/melatonin. Numerous studies have shown elevated levels of OS in pediatrics with ADHD, including high levels of urinary 8-hydroxy-2'deoxyguanosine (8-OHdG), plasma malondialdehyde (MDA), total oxidant status (TOS), oxidative stress index (OSI), and high activity of serum oxidative stress-inducing enzymes such as nitric oxide synthase (NOS) and xanthine oxidase (XO).

According to a previous study, the hyperactivity score on Conners' Teacher Rating Scale increased in correlation with increasing NOS enzyme activity, which can lead to progressive damage to the vulnerable pathways of attention and physical activity due to the production of NO radicals. Decreased antioxidant levels have been observed in pediatrics with ADHD, including low total antioxidant status (TAS), low activity of antioxidant enzymes such as glutathione S-transferase (GST) and paraxonase-1, glutathione peroxidase (GPx), and low serum total antioxidant capacity (TAC).

Neuroinflammation, along with OS, can activate astrocytes and microglia, leading to proinflammatory cytokine secretion and catecholaminergic dysregulation, which can exacerbate ADHD symptoms. Furthermore, inflammatory cytokines that can be released in response to psychological stress might interfere with the maturation of PFC and neurotransmitters implicated in ADHD. Pediatrics with ADHD exhibit elevated levels of inflammatory markers, including plasma C-reactive protein (CRP), IL-6, TNF-α and high activity of serum adenosine deaminase, an enzyme that increases in inflammatory diseases. An association between symptoms in children with ADHD and serum cytokines was seen in the elevation of IL-16 with hyperactivity and IL-13 with inattention.

Several treatment strategies are used for ADHD, including pharmacological, non-pharmacological or a combination of both, with pharmacological treatment being the mainstay, involving stimulants (methylphenidate, amphetamines) and non-stimulants (atomoxetine, guanfacine, clonidine).

Despite numerous studies on their efficacy and safety, these agents may not always be promising, as a proportion of patients may not respond or may not be able to tolerate their adverse events. Thus, increasing studies are exploring alternative therapies for ADHD, focusing on the neuroprotective effects of dietary and natural compounds like antioxidants that can be serving as an alternative or supplement to classical treatment with fewer side effects.

Research on antioxidants in pediatrics with ADHD has shown promising results in improving symptoms and reducing scores on ADHD questionnaires, as observed in Coenzyme Q10, Resveratrol, Vitamin D, L-carnosine, Ginkgo biloba, n-3 fatty acids, Pycnogenol, and Flax oil with vitamin C.

Nigella sativa (NS), Ranunculaceae family, is a highly valued nutraceutical herbal plant known as black seeds or black cumin. For centuries, people all around the world have utilized the seeds and oil of Nigella sativa to cure a broad range of illnesses. Nigella sativa seed, particularly its essential oil, contains thymoquinone, thymohydroquinone, thymol, carvacrol, nigellidine, nigellicine, and α-hederin. Thymoquinone (TQ) possesses the majority of nigella sativa oil (NSO) therapeutic benefits. Thymoquinone can be regarded as a useful substance targeting the central nervous system owing to its low molecular weight and lipophilic nature, which enable it to cross the blood-brain barrier.

Black seed oil (BSO) has shown anti-inflammatory and antioxidant properties in several human studies. Black seed oil supplementation significantly increased GPx in a previous human study.

Numerous in-vitro studies have shown that NS possesses neuroprotective effects that are attributed to its antioxidant and anti-inflammatory effects. Treatment with TQ significantly reduced neuronal cell death in the hippocampus, healed neural cells by increasing neural density after traumatic brain injury (TBI), and showed protective effects on neuronal nuclei and mitochondrial membranes by reducing MDA levels. Additionally, superoxide dismutase (SOD), GSH, and catalase activities were restored to normal levels with a reduction in lipid peroxidation. Thymoquinone significantly reduced inflammation, oxidative stress, neuronal cell death, and brain damage following ischemic stroke by targeting antioxidant pathways such as nuclear erythroid-2-related protein and heme-oxygenase-1 (Nrf2/HO-1).

Thymoquinone improved symptoms in a Parkinson disease (PD) rat model by preventing changes in dopamine levels in the substantia nigra. In a PD rat model, thymoquinone neuroprotection is partially attributed to the attenuation of lipid peroxidation, as seen in lowering MDA levels.

Previous human studies suggested that NS can stabilize mood, reduce anxiety, and regulate cognition, attention, and memory.

In rats, TQ administration significantly improved cognition by enhancing cholinergic function, synaptic plasticity, and attenuating oxidative damage and neuroinflammation, as shown by increased SOD and TAC and reduced MDA, NO, TNF-α immunoreactivity, and AChE activities. Thymoquinone also showed significant antianxiety-like activity in mice through possible modulation of NO and γ-aminobutyric acid (GABA) pathways. Clinically, Nigella sativa oil could enhance rats abilities of learning and memory.

In 2020, Folarin and his colleagues conducted an animal study to investigate the curative roles of Nigella sativa on the PFC functions of ADHD rat model. The nigella sativa followed by ethanol (NSE) mice group showed reduced inattentiveness and hyperactivity with lower levels of the excitatory neurotransmitter glutamate, and also showed higher recognition memory, antioxidant GPx levels, dopamine levels, and higher neuronal density compared to the ethanol group. These results suggest the protective effects of NS on PFC functions in ADHD mice model following maternal exposure to ethanol.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 12 years old who can swallow capsules.
* Diagnosed with ADHD according to the DSM-V criteria
* Having a stable dose of atomoxetine for at least 12 weeks prior to the study.

Exclusion Criteria:

* If there is any alteration in the ADHD treatment plan or being incompliant.
* Having any other psychiatric or neurological disorder that may interfere with the study outcomes like Autism, Anxiety, Obsessive compulsive disorder.
* Having any known allergy or hypersensitivity to black seed oil or its components.
* Having bleeding disorders or taking blood thinners.
* Having diabetes or taking medications that affect blood sugar levels.
* Having renal or hepatic impairment

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Serum Glutathione Perioxidase | 3 months
  Blood samples will be withdrawn from each patient at baseline and after 12 weeks. Samples will be centrifuged, and the sera will be separated and stored at -80°C till analysis. Serum GPx will be measured using human GPx ELISA kit at baseline and after 12 weeks.

SECONDARY OUTCOMES:
NICHQ Vanderbilt Assessment Scale-PARENT Informant | 3 months
  The symptoms and severity of ADHD will be assessed using NICHQ Vanderbilt Assessment Scale-PARENT Informant for children aged 6-12 at baseline and after 12 weeks.
  The initial assessment scale has a total of 55 items in two components: symptom assessment and impairment in performance. Symptom assessment screens for symptoms that meet criteria for both inattentive (1-9) and hyperactive (10-18) ADHD. Also screens for symptoms of three other co-morbidities: oppositional defiant (19-26), conduct (27-40), and anxiety/depression (41-47). A positive response in symptom screens is a 2 or 3 (often, very often).
  The second section of the scale has a set of performance measures (48-55), scored 1 to 5, with 4 and 5 being somewhat of a problem/problematic.
  To meet the DSM-5 criteria for ADHD diagnosis, one must score 2 or 3 on at least 6 out of either the inattentive 9 or hyperactive 9 core symptoms or both and score 4 or 5 on any of the performance questions.
Child Health Questionnaire Parent Form 28 item (CHQ-PF28) | 3 months
  To assess the impact of ADHD on quality of life, Child Health Questionnaire Parent Form 28 item (CHQ-PF28) will be completed by parents at baseline and after 12 weeks.
  The CHQ-PF28 measures the following scales: Physical Functioning (3 items), Role functioning: emotional/behavior (1 item), Role functioning: physical (1 item), Bodily Pain (1 item), General Behavior (4 items), Mental Health (3 items), Self Esteem (3 items), General Health (4 items), Change in Health (1 item), Parental Impact-Emotional (2 items), Parental Impact-Time (2 items), Family Activities (2 items), and Family Cohesion (1 item).
  Response options vary from four to six levels for the scales. Per scale, the items are summed up and transformed into a scale from 0 (worst possible score) to 100 (best possible score), yielding two summary component scores of physical (PhS) and psychosocial (PsS) health.

IPD SHARING:
Plan to Share IPD: No